CLINICAL TRIAL: NCT05886751
Title: Randomized Trial of Trust in Online Videos About Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20-00540
Record Dates: First submitted 2023-05-24; First posted 2023-06-02 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Prostate Cancer
Keywords: Trust
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Video About Screening with Black Doctor (Experimental)
  Interventions: Other: Black Doctor Screening Video
- Video About Screening with White Doctor (Experimental)
  Interventions: Other: White Doctor Screening Video
- Video About Screening with Black Patient (Experimental)
  Interventions: Other: Black Patient Screening Video
- Video About Screening with White Patient (Experimental)
  Interventions: Other: White Patient Screening Video
- Video about Clinical Trials with Black Doctor (Experimental)
  Interventions: Other: Black Doctor Clinical Trials Video
- Video about Clinical Trials with White Doctor (Experimental)
  Interventions: Other: White Doctor Clinical Trials Video
- Video about Clinical Trials with Black Patient (Experimental)
  Interventions: Other: Black Patient Clinical Trials Video
- Video about Clinical Trials with White Patient (Experimental)
  Interventions: Other: White Patient Clinical Trials Video

INTERVENTIONS:
Other: Black Doctor Screening Video — Participants will view an online video with a Black doctor speaking about prostate cancer screening.
  Arms: Video About Screening with Black Doctor
Other: White Doctor Screening Video — Participants will view an online video with a White doctor speaking about prostate cancer screening.
  Arms: Video About Screening with White Doctor
Other: Black Patient Screening Video — Participants will view an online video with a Black patient speaking about prostate cancer screening.
  Arms: Video About Screening with Black Patient
Other: White Patient Screening Video — Participants will view an online video with a White patient speaking about prostate cancer screening.
  Arms: Video About Screening with White Patient
Other: Black Doctor Clinical Trials Video — Participants will view an online video with a Black doctor speaking about prostate cancer clinical trials.
  Arms: Video about Clinical Trials with Black Doctor
Other: White Doctor Clinical Trials Video — Participants will view an online video with a White doctor speaking about prostate cancer clinical trials.
  Arms: Video about Clinical Trials with White Doctor
Other: Black Patient Clinical Trials Video — Participants will view an online video with a Black patient speaking about prostate cancer clinical trials.
  Arms: Video about Clinical Trials with Black Patient
Other: White Patient Clinical Trials Video — Participants will view an online video with a White patient speaking about prostate cancer clinical trials.
  Arms: Video about Clinical Trials with White Patient

SUMMARY:
The study team will evaluate the impact of video characteristics on health consumers' trust in online videos. Participants will be randomized to watch a video by one of four speakers about prostate cancer screening or clinical trials and complete a questionnaire (approximately 15 minutes total).

ELIGIBILITY:
Inclusion Criteria:

1. US adult age 40+
2. Enrolled in Dynata online survey panel

Exclusion Criteria:

1. Children
2. Individuals living outside the U.S.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3649 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2022-01-07 (Actual)

PRIMARY OUTCOMES:
Level of Trust in the Video | Visit 1 (Day 1)
  Trust will be reported as a score on a Likert scale and asked as the following question: How much do you trust the information in the video? The total range of score is 1-4, where (1) trust the information completely, (2) trust most of the information, (3) trust some of the information, (4) do not trust the information

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Loeb, MD, MSc, PhD(hc), Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data needed for the proposed biomedical research use according to data use agreement from both parties will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data after signing a data use agreement will have access to the data upon reasonable request for biomedical research purposes. Requests should be directed to stacy.loeb@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Result] Loeb S, Ravenell JE, Gomez SL, Borno HT, Siu K, Sanchez Nolasco T, Byrne N, Wilson G, Griffith DM, Crocker R, Sherman R, Washington SL 3rd, Langford AT. The Effect of Racial Concordance on Patient Trust in Online Videos About Prostate Cancer: A Randomized Clinical Trial. JAMA Netw Open. 2023 Jul 3;6(7):e2324395. doi: 10.1001/jamanetworkopen.2023.24395. PMID 37466938

DOCUMENTS (1):
  • Informed Consent Form (2022-05-12): https://cdn.clinicaltrials.gov/large-docs/51/NCT05886751/ICF_000.pdf